CLINICAL TRIAL: NCT01145170
Title: Use of Nimotuzumab and Radiotherapy in the Treatment of Pediatric Patients With Diffuse Intrinsic Brainstem Glioma
Brief Title: Nimotuzumab and Radiotherapy in Pediatric Patients With Glioma
Acronym: POLARIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Collaborators: Centro de Immunologia Molecular, Cuba (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF090
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2012-01

CONDITIONS: Diffuse Intrinsic Brainstem Gliomas
Keywords: brainstem gliomas; pediatric patients
MeSH Terms: interventions — Radiotherapy; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nimotuzumab (Experimental): The study consists of a single treatment group, which will receive the first-line therapy for the disease. The therapy is the standard radiotherapy and a dose of the investigational product (nimotuzumab) at 150 mg/m2.
  Interventions: Radiation: Radiotherapy; Biological: Nimotuzumab

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy will be given at the standard dose between 54 and 60 Gy for irradiation of tumors of the central nervous system.
Biological: Nimotuzumab — The patients will receive the induction therapy for 12 weeks. If the patient reaches a complete, partial response (CR, PR) to the treatment or is at least evaluated as stable disease (SD) on week 12, the consolidation therapy should be initiated. The consolidation therapy will consist of the nimotuzumab administration, every 2 weeks.

SUMMARY:
The study consists in only one treatment group, which will receive the first-line therapy for the disease - standard radiotherapy and a 150 mg/m2 dose of the investigational product (nimotuzumab)

DETAILED DESCRIPTION:
General Purpose

1. To determine the therapeutic efficacy of the treatment with nimotuzumab in combination with radiotherapy in pediatric patients with diffuse intrinsic astrocytic of the brainstem glioma

Specific Purposes

1. To determine the efficacy regarding the event-free survival (EFS) rate by 6 months of treatment.
2. To determine the overall survival time of the patients with diffuse intrinsic astrocytic tumors of the cerebral trunk treated with combined radiotherapy and nimotuzumab.
3. To determine the antitumoral objective response of the patients treated with combined radiotherapy and nimotuzumab.
4. To determine the duration time of the response in the cases of objective response reached (CR or PR) or disease stabilization.
5. To assess the toxicity of the combination AcM h-R3-nimotuzumab and radiotherapy in the patients enrolled in the clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients with diffuse intrinsic brainstem gliomas, documented by standard imaging techniques (MRI). Note: Tumor biopsy and histological confirmation are not required in this study.
2. Patients eligible for radiotherapy with Cobalt60. The patients should not have received a previous specific oncological treatment.
3. Aged > 3 years old < 18 years old
4. Patients with measurable lesions, defined as those that can be accurately measured in at least 2 dimensions (the 2 largest perpendicular diameters), using standard techniques (MRI).
5. Female patients with childbearing potential should present a negative pregnancy test and adopt effective birth control methods, in case they are sexually active.
6. Male patients who can father a child should adopt effective birth control methods, in case they are sexually active.
7. Life expectancy > 12 weeks
8. Health general status, according to Karnofsky Index > 40% (Karnofsky Index for patients > 16 years old), Lansky > 40% (for patients < 16 years old)
9. Laboratory parameters within the normal limits, defined as: Hematopoietic: Hemoglobin > 10 g/L, Total Leukocytes > 2 x 109 cells/L, Platelets > 100 x 109/L; Hepatic: Liver functioning within the normal limits and without hepatic diseases demonstrated by ALT, AST < 2.5 x above the reference value and Total Bilirubin < 1.5 x above the reference value; Renal function: Serum Creatinine < 1.5 x above the reference value.
10. The parents or legal guardians should express, voluntarily, in writing, that the patient will be enrolled in the study upon signature of the informed consent form. At the investigator's discretion, where applicable, the consent will be obtained from the minor.

Exclusion Criteria:

1. Low-grade brainstem glioma (e.g., focal, cervicomedullary, tectal brainstem glioma).
2. Patients previously treated with some AcM.
3. Patients previously treated with some antineoplastic therapy, including chemotherapy, immunotherapy or radiotherapy.
4. Concurrent treatment with some antineoplastic therapy not conceived in the study protocol.
5. Breastfeeding or pregnant patients.
6. Patients that, at the time of enrollment, have some related chronic disease under decompensation (e.g., cardiopathy, diabetes, hypertension).
7. Patients who have history of hypersensitivity to this or another similar product.
8. Fever, severe septic processes and/or severe or acute allergy.
9. Patients who are participating in another clinical study with therapeutic purposes for their disease based on the time of the study enrollment.
10. Presence of a second tumor.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Tumor Volume | 6 months
  A Magnetic Resonance Imaging (MRI) will be used for measuring the tumor volume and it will be performed before the enrollment in the clinical study and every 12 weeks. The patient follow-up will be performed for 2 years after his/her inclusion in the investigation. The final evaluation will be performed 2 years after the inclusion of the last patient.
  The main response variable will be the progression-free survival by 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sidnei Epelman, Principal Investigator — Casa de Saúde santa Marcelina; Vicente Odone Filho, Principal Investigator — Hospital das Clínicas da Faculda de Medicina da USP; Algemir L Brunetto, Principal Investigator — Hospital de Clínicas de Porto Alegre; Claudia T Oliveira, Principal Investigator — Hospital Amaral Carvalho
Locations (5):
- Brazil (4):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Casa de Saúde Santa Marcelina, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
- Hospital Juan Manuel Márquez, Havana, Cuba